CLINICAL TRIAL: NCT07320352
Title: Assessment of Changes in Labial Bone Thickness and Root Surface After Enmasse Retraction With and Without Hard Laser Assistance:Comparative Randomized Cllinical Trial
Brief Title: Assessment of Changes in Labial Bone Thickness and Root Surface After Enmasse Retraction With and Without Hard Laser Assistance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Faculty of Dental Medicine for Girls (Other Government)
Responsible Party: Principal Investigator, Salma Toubar, Principal investigator, Faculty of Dental Medicine for Girls
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ORTHO-108-2-K
Record Dates: First submitted 2025-11-23; First posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Amount of Labial Bone Thickness; Amount of Root Resorption

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enmass retraction with hard laser therapy and effect on labial bone thickness and root resorption (Experimental)
  Interventions: Procedure: Hard laser therapy biolase device
- Enmass retraction without hard laser therapy and effect on labial bone thickness and root resorption (Experimental)
  Interventions: Device: Enmass retraction without hard laser

INTERVENTIONS:
Procedure: Hard laser therapy biolase device — Enmass retraction after hard laser therapy with biolase machine
  Arms: Enmass retraction with hard laser therapy and effect on labial bone thickness and root resorption
Device: Enmass retraction without hard laser — with long hook and memory power chain
  Arms: Enmass retraction without hard laser therapy and effect on labial bone thickness and root resorption

SUMMARY:
Assessment of Changes in Labial Bone Thickness and Root Surface After Enmasse Retraction With and Without Hard Laser Assistance:Comparative Randomized Cllinical Trial

ELIGIBILITY:
Inclusion Criteria:

* class 2 division1 malocclusion
* Dentoalveolar bimaxillary protrusion
* Extraction of maxillary 1st premolars
* No evidence of root resorption
* cooperative patient

Exclusion Criteria:

* un cooperative patient
* Bleeding disorders

Ages: 16 Years to 23 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2024-02-28 (Actual); Primary Completion 2025-09-20 (Actual); Study Completion 2025-10-20 (Actual)

PRIMARY OUTCOMES:
evaluation of labial bone thickness with and without hard laser. | 1year
evaluation of root surface changes with and without hard laser. | 1year

CONTACTS AND LOCATIONS:
Locations (1):
- dental medicine of Al-Azhar university, girls branch., Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Almagrami I, Albarakani AY, Almashraqi AA, Alhammadi MS, Al-Warafi LA, Almaqrami M, Qiao Y. Volumetric and tridimensional root resorption and alveolar bone changes in Class II malocclusion extraction protocol treated with clear aligners and fixed orthodontic appliances: A comparative study. Am J Orthod Dentofacial Orthop. 2025 May;167(5):539-549. doi: 10.1016/j.ajodo.2024.11.012. Epub 2025 Jan 9. PMID 39797866
- See also: Volumetric and tridimensional root resorption and alveolar bone changes in Class II malocclusion extraction protocol — https://pubmed.ncbi.nlm.nih.gov/39797866/